CLINICAL TRIAL: NCT03623074
Title: Efficacy and Safety Study of Novel Spectacle Lens Designs to Control of Myopia
Brief Title: Control of Myopia Using Novel Spectacle Lens Designs
Acronym: CYPRESS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SightGlass Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPRO-1802-001
Record Dates: First submitted 2018-08-03; First posted 2018-08-09 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Juvenile Myopia
Keywords: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and parents of participants will be masked. Investigational site staff tasked with measuring key primary variables (i.e., axial length and SER) will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Test Arm 1 (Experimental): Single vision, impact-resistant spectacle lenses
  Interventions: Device: Novel spectacle lens design
- Test Arm 2 (Experimental): Single vision, impact-resistant spectacle lenses
  Interventions: Device: Novel spectacle lens design
- Test Arm 3 (Other): Single vision, impact-resistant spectacle lenses
  Interventions: Device: Spectacle lenses

INTERVENTIONS:
Device: Novel spectacle lens design — Use of lenses may reduce the rate of progression of juvenile myopia
  Arms: Test Arm 1; Test Arm 2
Device: Spectacle lenses — Use of lenses may reduce the rate of progression of juvenile myopia
  Arms: Test Arm 3

SUMMARY:
Randomized, controlled, multisite, subject-and observer-masked, 3-arm parallel group clinical trial of 36-month duration to evaluate the safety and efficacy of a novel spectacle lens design in reducing the progression of juvenile myopia.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-10 years of age (day prior to 10th birthday) at time of informed consent/assent
* SER error between -0.75 and -4.50 D
* SER power between the two eyes must be less than or equal to 1.50 D
* Willingness to participate in the trial for 3 years without content lens wear

Exclusion Criteria:

* Previous or current use of contact lenses
* Previous or current use of bifocals, progressive addition spectacles lenses
* Previous or current use of myopia control treatment
* Astigmatism worse then -1.25 DC in either eye

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 266 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Axial length | 36 Months
  Change in axial length from baseline
Spherical equivalent refraction | 36 Months
  Change in spherical equivalent refraction from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Rappon, OD, MS, FAAO, Study Chair — SightGlass Vision, Inc.
Locations (14):
- United States (13):
  - Golden Optometric Group, Whittier, California
  - Sabal Eye Care, Longwood, Florida
  - Visual Performance Center, Pensacola, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - Eye Associates of Northeast Louisiana (DBA Haik Humble Eye Center) Research Dept, West Monroe, Louisiana
  - Advanced Eyecare, PC, Raytown, Missouri
  - SUNY School of Optometry, New York, New York
  - Sacco Eye Group, Vestal, New York
  - Dept of Clinical Research, South Shore Eye Care, LLP, Wantagh, New York
  - Dunes Eye Consultants, Dakota Dunes, South Dakota
  - Total Eye Care, Memphis, Tennessee
  - University of Houston College of Optometry, Houston, Texas
  - William J Bogus, OD, FAAO, Salt Lake City, Utah
- Center for Ocular Research & Education, School of Optometry, University of Waterloo School of Optometry & Vision Science, Waterloo, Ontario, Canada

REFERENCES:
- [Derived] Rappon J, Chung C, Young G, Hunt C, Neitz J, Neitz M, Chalberg T. Control of myopia using diffusion optics spectacle lenses: 12-month results of a randomised controlled, efficacy and safety study (CYPRESS). Br J Ophthalmol. 2023 Nov;107(11):1709-1715. doi: 10.1136/bjo-2021-321005. Epub 2022 Sep 1. PMID 36126105